CLINICAL TRIAL: NCT03181503
Title: A Study to Assess the Safety and Efficacy of Nemolizumab (CD14152) in Subjects With Prurigo Nodularis (PN)
Brief Title: Safety and Efficacy of Nemolizumab in PN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.03.SPR.115828
Record Dates: First submitted 2017-06-07; First posted 2017-06-08 (Actual); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2019-11

CONDITIONS: Prurigo Nodularis
MeSH Terms: interventions — nemolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received 3 subcutaneous injections of placebo (matched to nemolizumab) every 4 weeks (Q4W) up to Week 8.
  Interventions: Drug: CD14152 placebo
- Nemolizumab 0.5 mg/kg (Experimental): Participants received 3 subcutaneous injections of nemolizumab 0.5 milligram per kilogram (mg/kg) Q4W up to Week 8.
  Interventions: Drug: CD14152 Dose A

INTERVENTIONS:
Drug: CD14152 Dose A — 3 subcutaneous injections (every 4 weeks during the 12-week treatment period)
  Other Names: Nemolizumab
  Arms: Nemolizumab 0.5 mg/kg
Drug: CD14152 placebo — 3 subcutaneous injections (every 4 weeks during the 12-week treatment period)
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to assess the safety and efficacy of nemolizumab in subjects with prurigo nodularis.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blinded, parallel group, multicenter study to evaluate the safety and efficacy of nemolizumab over a 12-week treatment period in patients suffering from prurigo nodularis compared to its placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of at least 18 years at screening
2. Clinical diagnosis of PN for at least 6 months with:

   * Prurigo lesions on upper limbs with or without lesions on the trunk or lower limbs
   * At least 20 nodules on the entire body with a bilateral distribution
3. Severe pruritus defined as follows on a Numerical Rating Scale (NRS)

   * At the Screening visit 1: Mean of the worst daily intensity of the NRS score is ≥ 7 over the previous 3 days
   * At the Baseline visit: Mean of the worst daily intensity of the NRS score is ≥ 7 over the previous week; NOTE: NRS score should be measured on at least 5 days during the week preceding the baseline visit.
4. Female subjects must fulfill one of the criteria below:

   * Female subjects of non-childbearing potential (postmenopausal [absence of menstrual bleeding for 1 year prior to screening, without any other medical reason], hysterectomy or bilateral oophorectomy);
   * Female subjects of childbearing potential who agree to a true abstinence (when in line with the preferred and usual lifestyle of the subject), or to use an effective method of contraception throughout the clinical trial and for 120 days after the last study drug administration:

Exclusion Criteria:

1. Chronic pruritus resulting from another condition than PN such as scabies, insect bite, lichen simplex chronicus, psoriasis, acne, folliculitis, habitual picking, lymphomatoid papulosis, chronic actinic dermatitis, dermatitis herpetiformis, sporotrichosis, bullous disease
2. Unilateral lesions of prurigo (e.g only one arm affected)
3. Cutaneous bacterial or viral infection within 1 week before the baseline visit.
4. Infection requiring treatment with oral or parenteral antibiotics, antivirals, antiparasitics or antifungals within 1 week before the screening visit, or during the screening period, unless completely resolved at the screening/ baseline visits respectively,
5. Any uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with the interpretation of the clinical trial results and/or put the subject at Chronic pruritus resulting from another condition than PN such as scabies, insect bite, lichen simplex chronicus, psoriasis, acne, folliculitis, habitual picking, lymphomatoid papulosis, chronic actinic dermatitis, dermatitis herpetiformis, sporotrichosis, bullous disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- LKH-Univ. Klinikum Graz, Graz, Austria
- France (4):
  - Centre-Hospitalier Universitaire (CHU) - Hopital Morvan - Br, Brest
  - CHU de Nice - Hôpital Archet 2, Nice
  - Hopital Saint-Louis - Dermatology, Paris
  - Centre Hospitalier Universitaire De Toulouse, Toulouse
- Germany (8):
  - Charite - Campus Charite Mitte (CCM) - Dermatologie & Allergologie - Dermatologie & Allergologie, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Klinikum der Johann-Wolfgang Goethe-Universität, Frankfurt
  - Unikl. Schleswig-Holstein - Lübeck, Lübeck
  - Universitätsmedizin Mainz, Mainz
  - Klinikum Der Universität München - Campus Innenstadt - Dermatologie und Allergologie, München
  - Universitätsklinikum Münster, Münster
  - Eberhard-Karls Universitaet Tuebingen - Universitaets Hautkl, Tübingen
- Poland (3):
  - Centrum Medyczne DERMED, Lodz
  - Dermoklinika Centrum Medyczne s.c. M.Kierstan, J.Narbutt, A.Lesiak, Lodz
  - Kliniczny Szpital Wojew. nr 1 im. F.Chopina w Rzeszowie, Rzeszów

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwatra SG, Rodriguez D, Dias-Barbosa C, Budhiarso I, Fofana F, Vernon M, Gabriel S, Piketty C, Puelles J. Validation of the Peak Pruritus Numerical Rating Scale as a Patient-Reported Outcome Measure in Prurigo Nodularis. Dermatol Ther (Heidelb). 2023 Oct;13(10):2403-2416. doi: 10.1007/s13555-023-00999-9. Epub 2023 Aug 24. PMID 37615836
- [Derived] Stander S, Yosipovitch G, Legat FJ, Lacour JP, Paul C, Narbutt J, Bieber T, Misery L, Wollenberg A, Reich A, Ahmad F, Piketty C. Trial of Nemolizumab in Moderate-to-Severe Prurigo Nodularis. N Engl J Med. 2020 Feb 20;382(8):706-716. doi: 10.1056/NEJMoa1908316. PMID 32074418

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 sites in 4 countries.
Pre-assignment Details: A total of 100 participants were screened, out of which 70 participants were randomized and treated (36 participants in Placebo and 34 participants in Nemolizumab group). Total 60 participants completed the study.
Groups:
- Placebo: Participants received 3 subcutaneous injections of placebo (matched to nemolizumab) every 4 weeks (Q4W) (at baseline, week 4 and week 8). Participants were further followed up for 6 weeks.
- Nemolizumab 0.5 mg/kg: Participants received 3 subcutaneous injections of 0.5 milligram per kilogram (mg/kg) of nemolizumab Q4W (at baseline, week 4 and week 8). Participants were further followed up for 6 weeks.
Period: Overall Study
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Started | 36 | 34
Treated | 36 | 34
Completed | 29 | 31
Not Completed | 7 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Placebo: Participants received 3 subcutaneous injections of placebo (matched to nemolizumab) Q4W (at baseline, week 4 and week 8). Participants were further followed up for 6 weeks.
- Nemolizumab 0.5 mg/kg: Participants received 3 subcutaneous injections of 0.5 mg/kg nemolizumab Q4W (at baseline, week 4 and week 8). Participants were further followed up for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (17.47) | 59.7 (13.16) | 56.0 (15.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 14 | 15 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 35 | 33 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Presence or absence of background of atopy [Count of Participants; unit: Participants]
  Presence | 6 | 5 | 11
  Absence | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Weekly Average of the Peak Pruritus Numeric Rating Scale (NRS) Score at Week 4 Using Last Observation Carried Forward (LOCF) Approach
Description: Pruritus NRS is a scale used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. Participants completed the assessment once daily at home in the evening. Participants were asked the following questions in their local language: 1) For average itch intensity: "on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable', how would you rate your itch overall during the previous 24 hours?"; 2) For maximum itch intensity: "on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Where, higher score indicated worst imaginable itch. Missing values including those who took rescue medication were replaced by LOCF approach.
Time Frame: Baseline, Week 4
Population: Intent-to-treat (ITT) population included all randomized participants and were analyzed 'as randomized' regardless of the treatment they received. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 34 | 33
Percent change | -13.8 (16.10) | -52.6 (33.96)

2. Primary Outcome: Percent Change From Baseline in Weekly Average of the Peak Pruritus Numeric Rating Scale Score at Week 4 Using Multiple Imputation (MI) Method
Description: Pruritus NRS is a scale used by the participants to report the intensity of their pruritus (itch) during the last 24. Participants completed the assessment once daily at home in the evening. Participants were asked the following questions in their local language: 1) For average itch intensity: "on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable', how would you rate your itch overall during the previous 24 hours?"; 2) For maximum itch intensity: "on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Where, higher score indicated worst imaginable itch. Multiple imputation generated twenty-five sets of data with missing values imputed from observed data using linear regression.
Time Frame: Baseline, Week 4
Population: ITT population included all randomized participants and were analyzed 'as randomized' regardless of the treatment they received.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 36 | 34
Percent change | -18.3 (22.39) | -52.0 (33.94)

3. Secondary Outcome: Percent Change From Baseline in Weekly Average of the Peak Pruritus Numeric Rating Scale Score at Each Visit Using LOCF Approach
Description: as for outcome 1
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 16 and 18
Population: ITT population included all randomized participants analyzed 'as randomized' regardless of the treatment they received. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants evaluable for each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 34 | 33
percent change
  Week 1: number analyzed (Participants) | 33 | 32
  Week 1 | -6.1 (11.45) | -26.0 (21.93)
  Week 2 | -7.4 (14.85) | -41.7 (30.31)
  Week 4 | -13.8 (16.10) | -52.6 (33.96)
  Week 8 | -19.7 (20.03) | -56.5 (34.73)
  Week 12 | -18.7 (22.80) | -61.8 (34.95)
  Week 16 | -20.8 (22.29) | -61.1 (35.35)
  Week 18 | -21.7 (22.95) | -59.6 (35.89)

4. Secondary Outcome: Absolute Change From Baseline in Weekly Average of the Peak Pruritus Numeric Rating Scale Score at Each Visit Using LOCF Approach
Description: as for outcome 1
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 16 and 18
Population: ITT population included all randomized participants analyzed 'as randomized' regardless of the treatment they received. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants evaluable at each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 34 | 33
Units on a scale
  Week 1: number analyzed (Participants) | 33 | 32
  Week 1 | -0.5 (0.87) | -2.1 (1.66)
  Week 2 | -0.6 (1.21) | -3.4 (2.38)
  Week 4 | -1.2 (1.33) | -4.3 (2.77)
  Week 8 | -1.6 (1.62) | -4.7 (2.90)
  Week 12 | -1.5 (1.84) | -5.1 (2.95)
  Week 16 | -1.7 (1.81) | -5.1 (3.00)
  Week 18 | -1.8 (1.87) | -4.9 (3.07)

5. Secondary Outcome: Percent Change From Baseline in Weekly Average of the Average Pruritus Numeric Rating Scale Score at Each Visit Using LOCF Approach
Description: Pruritus NRS is a scale used by the participants to report the intensity of their pruritus (itch) during the last 24. Participants completed the assessment once daily at home in the evening. Participants were asked the following questions in their local language: 1) For average itch intensity: "on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable', how would you rate your itch overall during the previous 24 hours?"; 2) For maximum itch intensity: "on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Where, higher score indicated worst imaginable itch. Missing values including those who took rescue medication were replaced by LOCF approach.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 16 and 18
Population: ITT population included all randomized participants and were analyzed 'as randomized' regardless of the treatment they received. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants evaluable for each time point.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 34 | 32
Percent change
  Week 1: number analyzed (Participants) | 33 | 31
  Week 1 | -7.5 (12.82) | -26.6 (21.25)
  Week 2 | -9.6 (15.28) | -44.0 (29.54)
  Week 4 | -16.5 (18.25) | -53.4 (33.23)
  Week 8 | -24.6 (23.38) | -57.3 (34.78)
  Week 12 | -23.0 (26.31) | -62.6 (34.98)
  Week 16 | -25.9 (24.89) | -62.4 (35.93)
  Week 18 | -26.2 (25.39) | -60.4 (36.15)

6. Secondary Outcome: Absolute Change From Baseline in Weekly Average of the Average Pruritus Numeric Rating Scale Score at Each Visit Using LOCF Approach
Description: as for outcome 1
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 16 and 18
Population: ITT population included all randomized participants and were analyzed 'as randomized' regardless of the treatment they received. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants evaluable at each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 34 | 32
Units on a scale
  Week 1: number analyzed (Participants) | 33 | 31
  Week 1 | -0.5 (0.82) | -1.9 (1.47)
  Week 2 | -0.8 (1.14) | -3.2 (2.03)
  Week 4 | -1.3 (1.41) | -3.9 (2.44)
  Week 8 | -1.9 (1.80) | -4.2 (2.60)
  Week 12 | -1.8 (2.05) | -4.6 (2.71)
  Week 16 | -2.0 (1.97) | -4.6 (2.86)
  Week 18 | -2.1 (2.02) | -4.5 (2.94)

7. Secondary Outcome: Percent Change From Baseline in Weekly Average of the Peak of Pruritus Verbal Rating Scale (VRS) Score at Each Visit Using LOCF Approach
Description: VRS consists of a list of adjectives describing different levels of symptom intensity used by participants to report intensity of their pruritus (itch) over last 24 hours. Participants marked on a 5-point VRS (0=no itch, 1=mild itch, 2=moderate itch, 3=severe itch, 4=very severe itch), a response that best described their pruritus intensity in last 24 hours. Participants were asked following questions in their local language: 1) For average itch intensity: "on a scale of 0-4, with 0 being 'no itch' and 4 being 'very severe itch', how would you rate your itch overall during previous 24 hours?"; 2) For maximum itch intensity: "on a scale of 0-4, with 0 being 'no itch' and 4 being 'very severe itch', how would you rate your worst itch during previous 24 hours?". Where, higher score indicated very severe itch. Missing values including those who took rescue medication were replaced by LOCF approach.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 16 and 18
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Nemolizumab 0.5 mg/kg: Participants received 3 subcutaneous injections of 0.5 mg/kg of nemolizumab Q4W (at baseline, week 4 and week 8). Participants were further followed up for 6 weeks.
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 34 | 32
Percent change
  Week 1: number analyzed (Participants) | 33 | 31
  Week 1 | -9.8 (14.24) | -27.6 (17.21)
  Week 2 | -12.3 (17.64) | -39.1 (25.38)
  Week 4 | -15.6 (20.95) | -50.7 (29.37)
  Week 8 | -20.7 (21.22) | -54.3 (30.61)
  Week 12 | -19.4 (23.60) | -56.9 (32.64)
  Week 16 | -21.2 (22.24) | -55.6 (34.48)
  Week 18 | -23.0 (21.97) | -53.4 (36.56)

8. Secondary Outcome: Absolute Change From Baseline in Weekly Average of the Peak of Pruritus Verbal Rating Scale Score at Each Visit Using LOCF Approach
Description: as for outcome 7
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12,16 and 18
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 34 | 32
Units on a scale
  Week 1: number analyzed (Participants) | 33 | 31
  Week 1 | -0.3 (0.47) | -0.9 (0.57)
  Week 2 | -0.4 (0.61) | -1.3 (0.83)
  Week 4 | -0.6 (0.74) | -1.6 (1.00)
  Week 8 | -0.7 (0.74) | -1.8 (1.06)
  Week 12 | -0.7 (0.83) | -1.8 (1.09)
  Week 16 | -0.7 (0.78) | -1.8 (1.16)
  Week 18 | -0.8 (0.77) | -1.7 (1.26)

9. Secondary Outcome: Percent Change From Baseline in Weekly Average of the Average Pruritus Verbal Rating Scale Score at Each Visit Using LOCF Approach
Description: as for outcome 7
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 16 and 18
Population: ITT population that included all randomized participants and were analyzed 'as randomized' regardless of the treatment they received. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants evaluable at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 34 | 32
percent change
  Week 1: number analyzed (Participants) | 33 | 31
  Week 1 | -10.5 (19.72) | -29.6 (16.90)
  Week 2 | -13.0 (19.20) | -42.9 (24.22)
  Week 4 | -16.4 (24.10) | -52.1 (27.63)
  Week 8 | -23.5 (22.89) | -55.4 (30.63)
  Week 12 | -21.9 (25.90) | -62.1 (29.98)
  Week 16 | -25.1 (24.15) | -62.0 (32.48)
  Week 18 | -26.2 (24.40) | -58.7 (34.81)

10. Secondary Outcome: Absolute Change From Baseline in Weekly Average of the Average Verbal Rating Scale Score at Each Visit Using LOCF Approach
Description: as for outcome 7
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12,16 and 18
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 34 | 32
Units on a scale
  Week 1: number analyzed (Participants) | 33 | 31
  Week 1 | -0.4 (0.50) | -0.9 (0.49)
  Week 2 | -0.4 (0.61) | -1.3 (0.68)
  Week 4 | -0.6 (0.73) | -1.6 (0.84)
  Week 8 | -0.7 (0.72) | -1.7 (0.96)
  Week 12 | -0.7 (0.82) | -1.9 (0.94)
  Week 16 | -0.8 (0.78) | -1.9 (1.06)
  Week 18 | -0.8 (0.79) | -1.8 (1.16)

11. Secondary Outcome: Dynamic Pruritus Score (DPS) at 24, 48, and 72 Hours After First Injection and Before Second Injection (Week 4)
Description: The 9-point DPS is a dynamic scale used by participants to evaluate the change of their pruritus compared with an earlier time point. The scale ranges from 0 (strongly worsened pruritus) to 8 ([almost] no pruritus anymore), including intermediate marks for slightly improved/worsened, moderately improved/worsened, and rather improved/worsened. Participants recorded their DPS score in their local language, and completed the assessment 24, 48 and 72 hours after the first injection at baseline and at week 4 before the second injection.
Time Frame: After 24, 48, 72 hours of first Injection and before second injection (Week 4)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 30 | 32
Units on a scale
  First injection, after 24 hours: number analyzed (Participants) | 23 | 22
  First injection, after 24 hours | 4.3 (0.96) | 5.0 (1.20)
  First injection, after 48 hours: number analyzed (Participants) | 22 | 23
  First injection, after 48 hours | 4.0 (1.69) | 5.3 (1.40)
  First injection, after 72 hours: number analyzed (Participants) | 25 | 24
  First injection, after 72 hours | 4.0 (1.37) | 5.7 (1.34)
  Before Second Injection (Week 4) | 4.4 (1.07) | 6.3 (1.89)

12. Secondary Outcome: Prurigo Activity Score (PAS) Item 5: Overall Number of Prurigo Lesions at Week 12
Description: PAS includes 7-descriptive items; 1) lesions type (papules nodules/plaques/umbilicated ulcers/ulcers/hypo-/hyperpigmented maculae); 2) number (prurigo lesions on whole body); 3) distribution (disseminated/localized [only 1/2 areas affected]/neither of them); 4) affected areas (forearm/upper arm/lower and upper leg/trunk/head); 5) number of prurigo lesions in selected area; 6) activity (prurigo lesions with excoriations/crusts and healed prurigo lesions compared to all prurigo lesions) and 7) front and back, areas of marked monitor lesions to recognize on next visit.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Prurigo Lesions
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 36 | 34
Prurigo Lesions
  Baseline | 87.1 (5.42) | 84.9 (5.50)
  Week 12 | 74.2 (6.83) | 54.8 (6.42)

13. Secondary Outcome: Prurigo Activity Score (PAS) Item 6: Number of Participants With Defined Stages of Excoriation/Crusts and Healed Lesions at Each Visit
Description: PAS includes 7-descriptive items; 1) lesions type (papules nodules/plaques/umbilicated ulcers/ulcers/hypo-/hyperpigmented maculae); 2) number (prurigo lesions on whole body); 3) distribution (disseminated/localized [only 1/2 areas affected]/neither of them); 4) affected areas (forearm/upper arm/lower and upper leg/trunk/head); 5) number of prurigo lesions in selected area; 6) activity (prurigo lesions with excoriations/crusts and healed prurigo lesions compared to all prurigo lesions) and 7) front and back, areas of marked monitor lesions to recognize on next visit. Item 6 has 5 stages (0-4) where each stage represents percentage of prurigo lesions with excoriations/crusts and healed prurigo lesions compared to all prurigo lesions: excoriations/crusts lesions; stage 0=0%, 1=1-25%, 2=26-50%, 3=51-75%, 4=76-100%; for healed lesions; stage 0=100%, 1=75-99%, 2=50-74%, 3=25-49%, 4=0-24%.
Time Frame: Day 1 (Baseline), Weeks 4, 8, 12 and 18
Population: ITT population included all randomized participants and were analyzed 'as randomized' regardless of the treatment they received. Here 'n' (number analyzed) signifies number of participants evaluable at each time point for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 36 | 34
Participants
  Excoriation/Crusts: Day 1: Stage 0 | 0 | 0
  Excoriation/Crusts: Day 1: Stage 1 | 2 | 4
  Excoriation/Crusts: Day 1: Stage 2 | 7 | 5
  Excoriation/Crusts: Day 1: Stage 3 | 14 | 12
  Excoriation/Crusts: Day 1: Stage 4 | 13 | 13
  Excoriation/Crusts: Week 4: Stage 0: number analyzed (Participants) | 34 | 33
  Excoriation/Crusts: Week 4: Stage 0 | 2 | 2
  Excoriation/Crusts: Week 4: Stage 1: number analyzed (Participants) | 34 | 33
  Excoriation/Crusts: Week 4: Stage 1 | 6 | 10
  Excoriation/Crusts: Week 4: Stage 2: number analyzed (Participants) | 34 | 33
  Excoriation/Crusts: Week 4: Stage 2 | 7 | 9
  Excoriation/Crusts: Week 4: Stage 3: number analyzed (Participants) | 34 | 33
  Excoriation/Crusts: Week 4: Stage 3 | 10 | 9
  Excoriation/Crusts: Week 4: Stage 4: number analyzed (Participants) | 34 | 33
  Excoriation/Crusts: Week 4: Stage 4 | 9 | 3
  Excoriation/Crusts: Week 8: Stage 0: number analyzed (Participants) | 32 | 32
  Excoriation/Crusts: Week 8: Stage 0 | 2 | 4
  Excoriation/Crusts: Week 8: Stage 1: number analyzed (Participants) | 32 | 32
  Excoriation/Crusts: Week 8: Stage 1 | 5 | 13
  Excoriation/Crusts: Week 8: Stage 2: number analyzed (Participants) | 32 | 32
  Excoriation/Crusts: Week 8: Stage 2 | 7 | 6
  Excoriation/Crusts: Week 8: Stage 3: number analyzed (Participants) | 32 | 32
  Excoriation/Crusts: Week 8: Stage 3 | 11 | 9
  Excoriation/Crusts: Week 8: Stage 4: number analyzed (Participants) | 32 | 32
  Excoriation/Crusts: Week 8: Stage 4 | 7 | 0
  Excoriation/CrustsWeek 12: Stage 0: number analyzed (Participants) | 30 | 32
  Excoriation/CrustsWeek 12: Stage 0 | 1 | 3
  Excoriation/Crusts: Week 12: Stage 1: number analyzed (Participants) | 30 | 32
  Excoriation/Crusts: Week 12: Stage 1 | 7 | 17
  Excoriation/Crusts: Week 12: Stage 2: number analyzed (Participants) | 30 | 32
  Excoriation/Crusts: Week 12: Stage 2 | 5 | 9
  Excoriation/Crusts: Week 12: Stage 3: number analyzed (Participants) | 30 | 32
  Excoriation/Crusts: Week 12: Stage 3 | 12 | 3
  Excoriation/Crusts: Week 12: Stage 4: number analyzed (Participants) | 30 | 32
  Excoriation/Crusts: Week 12: Stage 4 | 5 | 0
  Excoriation/Crusts: Week 18: Stage 0: number analyzed (Participants) | 30 | 31
  Excoriation/Crusts: Week 18: Stage 0 | 1 | 6
  Excoriation/Crusts: Week 18: Stage 1: number analyzed (Participants) | 30 | 31
  Excoriation/Crusts: Week 18: Stage 1 | 4 | 12
  Excoriation/Crusts: Week 18: Stage 2: number analyzed (Participants) | 30 | 31
  Excoriation/Crusts: Week 18: Stage 2 | 8 | 4
  Excoriation/Crusts: Week 18: Stage 3: number analyzed (Participants) | 30 | 31
  Excoriation/Crusts: Week 18: Stage 3 | 11 | 5
  Excoriation/Crusts: Week 18: Stage 4: number analyzed (Participants) | 30 | 31
  Excoriation/Crusts: Week 18: Stage 4 | 6 | 4
  Healed Lesions: Day 1: Stage 0 | 1 | 0
  Healed Lesions: Day 1: Stage 1 | 0 | 1
  Healed Lesions: Day 1: Stage 2 | 3 | 5
  Healed Lesions: Day 1: Stage 3 | 13 | 9
  Healed Lesions: Day 1: Stage 4 | 19 | 19
  Healed Lesions: Week 4: Stage 0: number analyzed (Participants) | 34 | 33
  Healed Lesions: Week 4: Stage 0 | 2 | 3
  Healed Lesions: Week 4: Stage 1: number analyzed (Participants) | 34 | 33
  Healed Lesions: Week 4: Stage 1 | 2 | 5
  Healed Lesions: Week 4: Stage 2: number analyzed (Participants) | 34 | 33
  Healed Lesions: Week 4: Stage 2 | 6 | 5
  Healed Lesions: Week 4: Stage 3: number analyzed (Participants) | 34 | 33
  Healed Lesions: Week 4: Stage 3 | 11 | 14
  Healed Lesions: Week 4: Stage 4: number analyzed (Participants) | 34 | 33
  Healed Lesions: Week 4: Stage 4 | 13 | 6
  Healed Lesions: Week 8: Stage 0: number analyzed (Participants) | 32 | 32
  Healed Lesions: Week 8: Stage 0 | 2 | 3
  Healed Lesions: Week 8: Stage 1: number analyzed (Participants) | 32 | 32
  Healed Lesions: Week 8: Stage 1 | 3 | 8
  Healed Lesions: Week 8: Stage 2: number analyzed (Participants) | 32 | 32
  Healed Lesions: Week 8: Stage 2 | 7 | 8
  Healed Lesions: Week 8: Stage 3: number analyzed (Participants) | 32 | 32
  Healed Lesions: Week 8: Stage 3 | 9 | 12
  Healed Lesions: Week 8: Stage 4: number analyzed (Participants) | 32 | 32
  Healed Lesions: Week 8: Stage 4 | 11 | 1
  Healed Lesions: Week 12: Stage 0: number analyzed (Participants) | 30 | 32
  Healed Lesions: Week 12: Stage 0 | 1 | 2
  Healed Lesions: Week 12: Stage 1: number analyzed (Participants) | 30 | 32
  Healed Lesions: Week 12: Stage 1 | 2 | 9
  Healed Lesions: Week 12: Stage 2: number analyzed (Participants) | 30 | 32
  Healed Lesions: Week 12: Stage 2 | 7 | 16
  Healed Lesions: Week 12: Stage 3: number analyzed (Participants) | 30 | 32
  Healed Lesions: Week 12: Stage 3 | 8 | 5
  Healed Lesions: Week 12: Stage 4: number analyzed (Participants) | 30 | 32
  Healed Lesions: Week 12: Stage 4 | 12 | 0
  Healed Lesions: Week 18: Stage 0: number analyzed (Participants) | 30 | 31
  Healed Lesions: Week 18: Stage 0 | 1 | 3
  Healed Lesions: Week 18: Stage 1: number analyzed (Participants) | 30 | 31
  Healed Lesions: Week 18: Stage 1 | 2 | 12
  Healed Lesions: Week 18: Stage 2: number analyzed (Participants) | 30 | 31
  Healed Lesions: Week 18: Stage 2 | 7 | 7
  Healed Lesions: Week 18: Stage 3: number analyzed (Participants) | 30 | 31
  Healed Lesions: Week 18: Stage 3 | 8 | 5
  Healed Lesions: Week 18: Stage 4: number analyzed (Participants) | 30 | 31
  Healed Lesions: Week 18: Stage 4 | 12 | 4

14. Secondary Outcome: Investigator Global Assessment (IGA) Score at Each Visit
Description: IGA is a 5-point scale used by the investigator or trained designee to evaluate the severity of the disease ranging from 0 to 4 where, 0 = clear, 1= almost clear, 2 = mild, 3 = moderate and 4 severe. IGA corresponds to the overall assessment of the severity of prurigo including presence of crust and nodules or skin bleeding. Higher score indicated greater severity of disease.
Time Frame: Day 1 (Baseline), Weeks 4, 8, 12 and 18
Population: ITT population included all randomized participants and were analyzed 'as randomized' regardless of the treatment they received. Here, 'n' (number analyzed) signifies number of participants evaluable for each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 36 | 34
Units on a scale
  Day 1 (Baseline) | 3.4 (0.49) | 3.5 (0.51)
  Week 4: number analyzed (Participants) | 35 | 33
  Week 4 | 3.3 (0.61) | 2.8 (0.81)
  Week 8: number analyzed (Participants) | 32 | 32
  Week 8 | 3.1 (0.67) | 2.4 (0.80)
  Week 12: number analyzed (Participants) | 30 | 32
  Week 12 | 2.8 (0.82) | 2.0 (0.80)
  Week 18: number analyzed (Participants) | 30 | 31
  Week 18 | 3.0 (0.93) | 2.0 (1.11)

15. Secondary Outcome: Percentage of Participants Achieving Investigator Global Assessment Success (Defined as IGA= 0 [Clear] or IGA = 1 [Almost Clear] With Two-point Improvement From Baseline) at Week 12
Description: as for outcome 14
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 36 | 34
percentage of participants | 2.8 | 20.6

16. Primary Outcome: Percent Change From Baseline in Weekly Average of the Peak Pruritus Numeric Rating Scale Score at Week 4 Using Observed Data
Description: Pruritus NRS is a scale used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. Participants completed the assessment once daily at home in the evening. Participants were asked the following questions in their local language: 1) For average itch intensity: "on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable', how would you rate your itch overall during the previous 24 hours?"; 2) For maximum itch intensity: "on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Where, higher score indicated worst imaginable itch.
Time Frame: Baseline, Week 4
Population: ITT population included all randomized participants and were analyzed 'as randomized' regardless of the treatment they received. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
Number analyzed (Participants) | 32 | 31
Percent change | -15.2 (17.42) | -54.9 (33.80)

ADVERSE EVENTS:
Time Frame: Up to 18 Weeks
Groups:
- Placebo: Participants received 3 subcutaneous injections of placebo (matched to nemolizumab) Q4W for 12 weeks (Baseline, Week 4 and Week 8). Participants were further followed up for 6 weeks.
- Nemolizumab 0.5 mg/kg: Participants received 3 subcutaneous injections of nemolizumab 0.5 mg/kg Q4W for 12 weeks (Baseline, Week 4 and Week 8). Participants were further followed up for 6 weeks.
Arm/Group | Placebo | Nemolizumab 0.5 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34
Serious Adverse Events (participants affected / at risk) | 3/36 | 4/34
Other Adverse Events (participants affected / at risk) | 22/36 | 26/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | Nemolizumab 0.5 mg/kg (N=34)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis Psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema Nummular (Skin and subcutaneous tissue disorders) | 0 | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Calculus Bladder (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | Nemolizumab 0.5 mg/kg (N=34)
Nasopharyngitis (Infections and infestations) | 4 | 5
Conjunctivitis (Infections and infestations) | 2 | 3
Bronchitis (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 2 | 0
Postoperative Wound Infection (Infections and infestations) | 2 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 5 | 2
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Increased Appetite (Metabolism and nutrition disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT03181503/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT03181503/SAP_001.pdf